CLINICAL TRIAL: NCT06706661
Title: Implementation of Nutritional Treatment to Older Patients Discharged With the Liaison Team
Brief Title: Implementation of Nutritional Efforts on Discharged Older Patients
Acronym: KMH2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Anne Marie Beck, Senior researcher, Herlev and Gentofte Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-24065575
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-04

CONDITIONS: Malnutrition
Keywords: food; dietician; malnutrition; nutrition risk; quality of life; muscle strength; readmissions; mortality; multimodal
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional treament (Experimental): At the day of discharge the intervention group (IG) receives a package containing foods and drinks covering dietary requirements for the next 24 h. Further, a goodie-bag containing samples of protein-rich milk-based drinks is provided. At day 4 after discharge, the IG receives dietetic counselling including a recommendation of daily exercise, and an individual nutrition plan. Information regarding recommendations of nutritional therapy after discharge is systematically and electronically communicated to the municipality. The dietician performes telephone follow-ups on day 30 and a home visit at 12 weeks
  Interventions: Other: Nutritional treatment

INTERVENTIONS:
Other: Nutritional treatment — At the day of discharge the intervention group (IG) receives a package containing foods and drinks covering dietary requirements for the next 24 h. Further, a goodie-bag containing samples of protein-rich milk-based drinks is provided. At day 4 after discharge, the IG receives dietetic counselling including a recommendation of daily exercise, and an individual nutrition plan. Information regarding recommendations of nutritional therapy after discharge is systematically and electronically communicated to the municipality. The dietician performes telephone follow-ups on day 30 and a home visit at 12 weeks

SUMMARY:
The aim of the study is to implement a nutritional treatment when discharging older patients at risk of malnutrition.

Data collected in the study will include an assessment of whether a combination of nutritional treatment and a liaison team reduces the risk of readmissions and mortality, improves nutritional status, physical function and quality of life

DETAILED DESCRIPTION:
During hospitalization, many older patients are at risk of malnutrition. Malnutrition in older adults is related to reduced physical function, more complications, re-admissions, days in hospital and reduced quality of life. As hospitalizations are often short (approximately 5 days), it is important to focus on nutritional intake during the convalescence period.

Upon discharge, a "Nutrition Gap" often occurs in practice, where the patient does not consume sufficient nutrition to ensure an optimal convalescence period. The lack of nutritional follow-up in connection with the discharge of older patients has been shown to have a markedly negative effect on, among other things, functional ability and readmissions. A study from Herlev Hospital, where the effect of a nutritional treatment upon discharge of older patients was investigated, showed a significant effect on muscle strength, quality of life and nutritional status. Another study from Herlev Hospital has shown that by associating a clinical dietitian with a liaison team and thus focusing on nutrition, the readmission rate was halved.

The problem is that it has not been investigated whether such a cross-sectoral effort can be implemented in practice and the results confirmed.

Hypothesis 1 is that it is possible to include and retain the older patients who are discharged with the liaison team for an effort that includes treatment of the risk of malnutrition and that the older participants find the effort relevant

Hypothesis 2 is that nutritional treatment will be able to reduce the number of unintended readmissions and thereby be cost-effective. Furthermore, it is expected that the nutritional treatment will increase the participants' nutritional status, muscle strength, muscle mass, quality of life and possibly have a positive effect on mortality.

ELIGIBILITY:
Inclusion Criteria:

Prescription of the Liaison team At nutritional risk according to NRS2002 Age 50+ Can read, hear and understand Danish or English Cognitive able to participate in the study, based on whether they are informed in time, place and own data

Exclusion Criteria:

Receives enteral or parenteral nutrition Following a special diet including texture modified food and drinks Short life expectancy Not deemed eligible by the project staff

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility | Assessed at baseline
  Eligibility will be assessed as the number of patients who fulfil the inclusion criteria out of the number of patients discharged with the liaison team
Recruitment | Assessed at baseline
  Recruitment rate will be assessed as the number of patients recruited out of the number of eligible patients
Retention | Assessed at three months
  Retention rate will be assessed as the number of patients who complete the nutritional treatment out of the total number of patients recruited

SECONDARY OUTCOMES:
Mortality | 30 days, 12 weeks, 6 monts, 1 year and 3 year
  health care records
Hospital re-admissions | 30 days, 12 weeks, 6 monts, 1 year and 3 year
  health care records
Health related Quality of life | 12 weeks
  Euro-qol tool EQ5D5L
Appetite | 30 days, 12 weeks
  SNAQ with a score from 5 to 20 where a score at or below 14 can predict weight loss
Muscle strenght | 4 days, 30 days, 12 weeks
  30 seconds chair stand
Dietary intake | 30 days, 12 weeks
  24 hours recall
weight | 4 days, 30 days
  body weight measurement
muscle mass | 12 weeks
  calf circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to GDPR

REFERENCES:
- [Result] Beck A, Andersen UT, Leedo E, Jensen LL, Martins K, Quvang M, Rask KO, Vedelspang A, Ronholt F. Does adding a dietician to the liaison team after discharge of geriatric patients improve nutritional outcome: a randomised controlled trial. Clin Rehabil. 2015 Nov;29(11):1117-28. doi: 10.1177/0269215514564700. Epub 2014 Dec 31. PMID 25552522
- [Result] Munk T, Svendsen JA, Knudsen AW, Ostergaard TB, Thomsen T, Olesen SS, Rasmussen HH, Beck AM. A multimodal nutritional intervention after discharge improves quality of life and physical function in older patients - a randomized controlled trial. Clin Nutr. 2021 Nov;40(11):5500-5510. doi: 10.1016/j.clnu.2021.09.029. Epub 2021 Sep 24. PMID 34656032